CLINICAL TRIAL: NCT02919644
Title: Vaccination with Autologous Dendritic Cells Loaded with Autologous Tumour Homogenate After Curative Resection for Stage IV Colorectal Cancer: a Phase II Study
Brief Title: Vaccination with Autologous Dendritic Cells Loaded with Autologous Tumour Homogenate After Curative Resection for Stage IV Colorectal Cancer.
Acronym: COREVAX-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST153.04; 2015-000894-11 (EudraCT Number)
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stage IV Colorectal Cancer; Curative Resection
Keywords: vaccination; autologous dendritic cells; autologous tumour homogenate; curative resection; stage IV colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vaccine + Interleukin -2 (IL2) (Experimental): autologous dendritic cells loaded with autologous tumour homogenate given by intradermal injection (day 1), followed by IL-2 given by subcutaneous injection daily for five days (days 3-7)
  Interventions: Biological: autologous dendritic cells loaded with autologous tumour homogenate; Drug: IL2

INTERVENTIONS:
Biological: autologous dendritic cells loaded with autologous tumour homogenate — Each vaccine dose consists of 10_7 autologous dendritic cells loaded with autologous tumor homogenate
Drug: IL2 — Each vaccine dose is followed, after two days, by IL-2 as adjuvant, at a dose of 3 MU daily for five consecutive days

SUMMARY:
Single-arm, monocentric trial to assess safety and immunological efficacy of adjuvant vaccination with autologous dendritic cells loaded with autologous tumour homogenate after curative resection for stage IV colorectal cancer

DETAILED DESCRIPTION:
Vaccination with autologous dendritic cells loaded with autologous tumour homogenate after curative resection for stage IV colorectal cancer: a phase II study.

Primary objectives: Safety Immunological efficacy, expressed as number of patients who show enhancement of the proportion of circulating immune effectors specific for a selected panel of Colon-Rectal Cancer (CRC)-associated antigens.

Secondary objectives: Clinical outcome of the patients (OS, RFS, TTR). To evaluate the predictive role of the development of a positive DTH test after at least three vaccine administrations.

To evaluate the persistence of an antitumor immune response after the completion of the vaccination program.

To evaluate the prognostic or predictive role of the enhancement of a specific immune response.

To evaluate a panel of inflammatory cytokines involved in antitumor immune response.

To evaluate the predictive role of immune cells in tumour microenvironment. To evaluate the predictive role of tumour antigen expression.

This is a two-stage, phase 2 clinical trial designed according to Simon minimax design. A 40% immune response rate would preclude further studies, while a 70% immune response rate would indicate that further studies would be warranted. Given α and β error of 0.1, the first stage will require enrolment of 7 patients. If at least 3 patients show an immune response and toxicity is acceptable, the study will proceed to the second stage and additional 12 patients will be enrolled.

The vaccine will be considered immunologically active if at least 11 patients are immunological responders.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed stage IV colorectal cancer surgically treated with radical intent.
2. The autologous surgical specimen must have been collected and sent to the Somatic Cell Therapy Lab of Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST IRCCS) and must fulfil all the acceptance criteria prescribed by the Good Manufacturing practise (GMP) procedures.
3. The patient must be disease-free, as assessed by CT scan or MRI of the chest, abdomen, pelvis performed within 60 days before enrolment. If the resected lesions had occurred in other sites, these must be also included in the baseline CT scan and in all the subsequent evaluations.
4. The patient must have recovered (grade 1 or less by CTCAE 4.0) from all the adverse events related to previous surgery.
5. Age >18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Patient must have acceptable organ function, defined as:

   1. Haemoglobin >10 g/dl
   2. White blood cells ≥4000/μl.
   3. Absolute neutrophil count >1500/μl.
   4. Platelets ≥100000/μl.
   5. aspartate aminotransferase (AST) and Alanine Aminotransferase (ALT) <3 times the upper institutional reference level.
   6. Total bilirubin <1.5 times the upper institutional reference level.
   7. Serum creatinine <1.5 times the upper institutional reference level.
8. Patients aged 70 years or older must have left ventricular ejection fraction not lower than 55% as assessed by echocardiography.
9. Female patients of childbearing potential and all male patients must accept and be compliant with an highly effective contraceptive method (i.e. with a failure rate of <1% per year: double barrier method, one barrier method plus spermicidal, intrauterine device, or oral contraception) from informed consent signature and up to three months after end of study. For this purpose are considered of childbearing potential all female subjects after puberty unless they are post-menopausal for at least two years or are surgically sterile. Complete abstinence from sexual intercourses is acceptable if patients' lifestyle guarantees his/her strict compliance with this prescription in the judgement of the Investigator.
10. The patient is willing and able to give written informed consent for the study.

Exclusion Criteria:

1. Patients with residual disease after surgery. Marginal resection of any lesion in the absence of clinically evident residual disease is acceptable.
2. Patients who relapsed within 6 months since primary treatment of stage I-III colorectal cancer. If adjuvant chemotherapy had been administered, the term must be computed since last chemotherapy dose.
3. Patient who completed surgery more than 60 days before study enrolment.
4. History of other neoplastic diseases in the previous 5 years, except basal cell carcinoma of the skin and in situ carcinoma of the cervix uteri treated with curative surgery.
5. History of congenital or acquired immunodeficiency, including history of organ transplantation.
6. Any positivity for the serologic markers of hepatitis B virus (HBV) (including at least anti-HBs antibodies and anti-hepatitis B core (HBc) antibodies), hepatitis C virus (HCV), HIV or Treponema pallidum. The serologic tests must have been performed within 30 days before any GMP-regulated activity (i.e. surgical resection and leukapheresis). The sole positivity for antibodies against the HBV S antigen (i.e. with all other HBV markers negative) is indicative of previous HBV vaccination and therefore is acceptable.
7. Female patients who are pregnant or nursing.
8. Patients undergone surgery after preoperatory chemotherapy with a fluoropyrimidine plus oxaliplatin, unless they are not candidate for postoperatory chemotherapy with the same schedule in the opinion of the Investigator (e.g. for unacceptable toxicity) or refuse completion of the perioperatory treatment.
9. Participation in another clinical trial with any investigational agent within 30 days prior to study screening.
10. Any active inflammatory or autoimmune disease requiring systemic steroids or other immunomodulatory agents as detailed in section 6.4, or potentially requiring such treatments during the study treatment in the judgement of the Investigator.
11. Any clinical condition that, in the opinion of the Investigator or the Transfusion Medicine specialist, is a contraindication to leukapheresis. In addition, all patients aged 70 or older must be evaluated by a cardiology specialist before the procedure to exclude any clinically relevant cardiac condition and any grade 3-4 cardiac arrhythmia, even if asymptomatic.
12. Any clinical condition that, in the opinion of the Investigator, contraindicates the subcutaneous administration of low-dose IL-2 as per protocol (see section 6.2 for details).
13. Any uncontrolled serious intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations potentially impacting patient safety and compliance in the opinion of the Investigator.
14. Refusal of giving written informed consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2016-12-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | up to 24 months
  To characterize the safety of the study drugs all adverse events observed during the study will be collected and assessed using the CTCAE v 4.03 criteria . Type, incidence, and severity of the adverse events will be reported and analyzed using descriptive statistics. All patients who received at least one treatment cycle will be considered evaluable for this primary endpoint.
immunological efficacy | up to 24 months
  Immunological efficacy will be assessed by quantifying circulating immune effectors specific for a selected panel of tumour antigens using interferon (IFN) - γELISPOT analysis . The assay determines the proportion of peptide-reactive T lymphocytes from peripheral blood mononuclear cells (PBMC) expressed as number of spot-forming Cells

SECONDARY OUTCOMES:
Relapse Free Survival (RFS) | up to 7 years
  Relapse Free Survival (RFS) is calculated as the time from study enrolment to either disease recurrence, defined as above, or the date of death for any cause. Patients alive with no evidence of disease recurrence at the time of their last visit are censored at the time of the last examination.
Overall Survival (OS) | up to 7 years
  Overall Survival (OS) is calculated as the time from study enrolment to the date of death for any cause. Patients still alive at the time of analysis are censored at the last time they are known to be alive.
Positive Delayed Type Hypersensitivity (DTH) skin test | up 24 months
  evaluation of the predictive role of a positive DTH test after at least three vaccine administrations
Antitumor Immune response | up to 7 years
  evaluation of the persistence of an antitumor immune response after the completion of the vaccination program assessed by ELISPOT assays
evaluation of the prognostic or predictive role of the enhancement of a specific immune response | up to 7 years
  evaluation of the prognostic or predictive role of the enhancement of a specific immune response assessed by ELISPOT
evaluation of a panel of inflammatory cytokines involved in antitumor immune response | up to 24 months
  Serum sampling will allow the evaluation of a panel of inflammatory cytokines during and after treatment and their concentration will be evaluated by SearchLight multiplex array analysis according to manufacturer's instructions (FDA-validated test)
evaluation of the predictive role of tumour antigen expression | up to 24 months
  Immunohistochemistry on formalin-fixed, paraffin-embedded tumour samples will allow to evaluate the expression of tumour-associated antigen
evaluation of the predictive role of immune cells in tumor microenvironment | up to 24 months
  Immunohistochemistry on formalin-fixed, paraffin-embedded tumour samples will allow to characterize the immune infiltrate

CONTACTS AND LOCATIONS:
Overall Officials: Francesco De Rosa, MD, Principal Investigator — UO Immunoterapia e Laboratorio TCS Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) S.r.l IRCCS
Locations (2):
- Italy (2):
  - UO Immunoterapia e Laboratorio TCS Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) S.r.l IRCCS, Meldola, FC
  - CRO-IRCCS Aviano, Aviano

IPD SHARING:
Plan to Share IPD: Undecided